CLINICAL TRIAL: NCT07002983
Title: Motor Control Retraining Exercises On Shoulder Dysfunction Post Mastectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Tarek Mohamed Hashem, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005751
Record Dates: First submitted 2025-05-19; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Post Mastectomy
Keywords: motor control; shoulder dysfunction; post mastectomy

STUDY DESIGN:
Intervention Model Description: the study will be 2 armed, single blind, parallel group, randomized controlled trial
Who Masked: Participant
Masking Description: single blind participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (motor control retraining group) (Active Comparator): This group will include 30 patients with post mastectomy shoulder dysfunction who will receive motor control retraining exercises in addition to their conventional physical therapy program, three sessions per week for 8 weeks, for 45:60 minutes according to patient's ability
  Interventions: Other: motor control retraining exercises; Other: traditional physical therapy for shoulder dysfunction
- control group ( conventional treatment group) (Placebo Comparator): This group will include 30 patients with post mastectomy shoulder dysfunction who will receive conventional physical therapy program in the form of shoulder joint mobilization, posterior capsule stretching and shoulder range of motion exercise (ROM) (Codman's pendulum exercises) for 30 minutes according to patient's ability, three sessions per week for 8 weeks
  Interventions: Other: traditional physical therapy for shoulder dysfunction

INTERVENTIONS:
Other: motor control retraining exercises — The motor control retraining package was targeted at correcting movement impairments of the scapula by re-educating muscle recruitment. There were two components to the package:
  1. Motor control exercises to correct alignment and coordination, which involve a) learning optimal scapular orientation at rest and then controlling optimal orientation during active arm movements; b) muscle specific exercises for trapezius and serratus anterior
  2. Manual therapy techniques commonly used in clinical practice to manage symptoms, as trigger point therapy and pectoralis minor supine manual stretch will be performed as necessary.
  Arms: study group (motor control retraining group)
Other: traditional physical therapy for shoulder dysfunction — shoulder joint mobilization, posterior capsule stretching and shoulder range of motion exercise (ROM) (Codman's pendulum exercises)
  Other Names: conventional treatment

SUMMARY:
Motor control and strengthening exercises can improve function in shoulder impingement patients by realigning the scapula and changing muscle recruitment patterns. Peripheral musculoskeletal impairments can be associated with cortical reorganisation. Movement retraining using the principles of motor control retrain muscle recruitment patterns and improve scapular kinematics, reducing subacromial impingement, thus improving function and reducing pain.

Furthermore, the need of this study is developed from the lack in the quantitative knowledge and information in the published studies about the effect of motor control retraining exercises on shoulder dysfunction post-mastectomy.

DETAILED DESCRIPTION:
sixty patients suffering from post-mastectomy shoulder dysfunction will participate in this study. Their ages will range from 40 to 55 years. The participants will be selected from Cairo university hospitals.

Design of the study:

In this randomised controlled trial study (RCT), the patients will be randomly assigned into two equal groups (30 patients for each group):

Group A (study group):

This group will include 30 patients with post mastectomy shoulder dysfunction who will receive motor control retraining exercises in addition to their conventional physical therapy program, three sessions per week for 8 weeks, for 45:60 minutes according to patient's ability.

Group B (control group):

This group will include 30 patients with post mastectomy shoulder dysfunction who will receive conventional physical therapy program in the form of shoulder joint mobilization, posterior capsule stretching and shoulder range of motion exercise (ROM) (Codman's pendulum exercises) for 30 minutes according to patient's ability, three sessions per week for 8 weeks.

Measurement equipment:

* Hand-held dynamometer: for measurement of muscle strength.
* Digital inclinometer: for measurement of shoulder flexion, abduction and scapular upward rotation.
* Shoulder Pain and Disability Index (SPADI): for measurement of shoulder disability.

Therapeutic procedures:

• Motor control retraining exercises of the scapular musculature.

Motor control retraining exercises:

The motor control retraining package was targeted at correcting movement impairments of the scapula by re-educating muscle recruitment. There were two components to the package:

1. Motor control exercises to correct alignment and coordination, which involve a) learning optimal scapular orientation at rest and then controlling optimal orientation during active arm movements; b) muscle specific exercises for trapezius and serratus anterior
2. Manual therapy techniques commonly used in clinical practice to manage symptoms, as trigger point therapy and pectoralis minor supine manual stretch will be performed as necessary.

   * Traditional physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* The subject selection will be according to the following criteria:

  * Female patients with age range between 40-55 years.
  * All patients have shoulder dysfunction.
  * Patients were 2 months to 4 months post modified radical mastectomy or axillary lymph node dissection.
  * Patients received their radiotherapy or chemotherapy or both.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:

  * Rheumatoid arthritis.
  * History of trauma or accidental injuries.
  * Neurological involvement (stroke, Parkinsonism).
  * History of surgery on involved shoulder.
  * Diabetic patient.
  * Moderate and severe lymphoedema.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females who have shoulder dysfunction post mastectomy
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Instrumented digital hand-held dynamometer | 8 weeks
  Hand-held dynamometry (Lafayette manual muscle tester) will be used to measure isometric strength of shoulder flexion and abduction. It is an ergonomic hand-held device for objectively providing reliable, accurate readings that conform to most manual muscle testing protocols. It has good to excellent validity and reliability for most measures of isometric muscle strength particularly for proximal muscle groups.
Digital inclinometer | 8 weeks
  A digital inclinometer is used to measure shoulder flexion, abduction and upward rotation of scapula. It has digital screen that display the angle at which the inclinometer is situated allowing direct joint angle measurements

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 8 weeks
  The SPADI is a self-administered questionnaire that contains thirteen items which assess two domains (pain and disability) (Shamley et al., 2012). It has an 8-item subscale to evaluate disability and a 5-item subscale to measure pain. Each subscale is summed and transformed to a score out of 100. A mean is taken of the two subscales to give a total score out of 100, higher score indicating greater impairment or disability

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Tarek, PhD, Principal Investigator — Teaching assistant physical therapy for surgery cairo university
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publication at international journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: january, 2027
Access Criteria: open access

DOCUMENTS (1):
  • Study Protocol (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT07002983/Prot_000.pdf